CLINICAL TRIAL: NCT02558036
Title: Optimal Head and Neck Position for Intubation During Videolaryngoscopy: Comparison Between "Sniffing" and Neutral Position Using Channelled and Non-channelled Videolaryngoscopes
Brief Title: Optimal Head and Neck Position During Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 178075
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Head and Neck Position for Intubation
Keywords: Head Neck Position Videolaryngoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C-Mac D-Blade Neutral Position (Active Comparator): C-Mac D-Blade videolaryngoscope with patients head and neck in neutral position.
  Interventions: Other: C-Mac D-Blade Videolaryngoscope
- C-Mac D-Blade Sniffing Position (Active Comparator): C-Mac D-Blade videolaryngoscope with patients head and neck in sniffing position.
  Interventions: Other: C-Mac D-Blade Videolaryngoscope
- King Vision Neutral Position (Active Comparator): King Vision videolaryngoscope with patients head and neck in neutral position.
  Interventions: Other: King Vision Videolaryngoscope
- King Vision Sniffing Position (Active Comparator): King Vision videolaryngoscope with patients head and neck in sniffing position.
  Interventions: Other: King Vision Videolaryngoscope

INTERVENTIONS:
Other: C-Mac D-Blade Videolaryngoscope — Using C-Mac D-Blade Videolaryngoscope patients will be positioned the neutral Head and Neck Position
  Arms: C-Mac D-Blade Neutral Position
Other: C-Mac D-Blade Videolaryngoscope — Using C-Mac D-Blade Videolaryngoscope patients will be positioned in Sniffing Head and Neck Position
  Arms: C-Mac D-Blade Sniffing Position
Other: King Vision Videolaryngoscope — Using the King Vision Videolaryngoscope patients will be positioned in the neutral Head and Neck Position
  Arms: King Vision Neutral Position
Other: King Vision Videolaryngoscope — Using the King Vision Videolaryngoscope patients will be positioned in Sniffing Head and Neck Position
  Arms: King Vision Sniffing Position

SUMMARY:
Optimal patient head and neck position when performing videolaryngoscopy for endotracheal intubation has not yet been established.The investigators aim to assess the effect of two different positions on the laryngeal view obtained and success of tracheal intubation during videolaryngoscopy with two commercially available and well established videolaryngoscopes.

DETAILED DESCRIPTION:
The optimum patient head and neck position for direct laryngoscopy (when the anaesthetist views the larynx with a curved metallic blade before passing a tube for ventilation of the lungs) is traditionally considered to be the "sniffing the morning air" (neck flexion and head extension) position. This has been questioned previously as there is no randomized controlled study to date to explore this statement. The patient should be optimally positioned prior to induction of anaesthesia, especially because in the event of an unexpected difficult intubation, the Difficult Airway Society guidelines suggest the use of an alternative laryngoscope. In current clinical practice a videolaryngoscope (a curved blade with a camera attached to it that allows the anaesthetist to see around corners) has been used as an alternative laryngoscope. To the best of our knowledge, the ideal patient position for videolaryngoscopy has not yet been described. The intubation time and rate of success at intubation using a C-Mac D-Blade videolaryngoscope was previously assessed by Serocki et al, but only in the sniffing position. It is possible that adopting a different position when using the C-Mac D- Blade might result in a superior view of the larynx. Furthermore, the optimal patient position has not yet been assessed for intubation with the King Vision videolaryngoscope.

This key information could gain precious seconds in a difficult airway scenario (when securing the airway with a tube for ventilation proves difficult) and has obvious implications for patient management. The answer to this question could also help the anaesthetists take informed decisions when using videolaryngoscopy to intubate the trachea in elective settings. The investigators aim to assess the effect of two different positions on the laryngeal view obtained during videolaryngoscopy with two commercially available and well established videolaryngoscopes to try and answer this question.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and above, presenting for elective surgical procedure and requiring tracheal intubation will be invited to take part in the study.

Exclusion Criteria:

* Patients who are refusing to take part, below 18 years of age, pregnant women, American society of anaesthesiologists' class 4 and above, those requiring rapid sequence indication, super morbidly obese (BMI >50) and those patients requiring awake fibreoptic intubation will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Optimal Head and Neck Position during Videolaryngoscopy | 6 months
  This will be assessed using a Difficult Intubation Scale Score for each of the 2 videolaryngoscopes used in the study, which will be assessed in both neutral and sniffing positions.

SECONDARY OUTCOMES:
Laryngoscopy Time | Less than 1 minute
  From when the laryngoscope enters the mouth until achieving the best view of the larynx.
Intubation Time | Less than 1 minute
  from entering the mouth with the videolaryngoscope until endotracheal tube is inserted in the wind-pipe and the capnography trace is first visible on the screen.

CONTACTS AND LOCATIONS:
Overall Officials: Cyprian Mendonca, Principal Investigator — Consultant
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El-Orbany M, Woehlck H, Salem MR. Head and neck position for direct laryngoscopy. Anesth Analg. 2011 Jul;113(1):103-9. doi: 10.1213/ANE.0b013e31821c7e9c. Epub 2011 May 19. PMID 21596871
- [Result] Adnet F, Baillard C, Borron SW, Denantes C, Lefebvre L, Galinski M, Martinez C, Cupa M, Lapostolle F. Randomized study comparing the "sniffing position" with simple head extension for laryngoscopic view in elective surgery patients. Anesthesiology. 2001 Oct;95(4):836-41. doi: 10.1097/00000542-200110000-00009. PMID 11605921
- [Result] Serocki G, Neumann T, Scharf E, Dorges V, Cavus E. Indirect videolaryngoscopy with C-MAC D-Blade and GlideScope: a randomized, controlled comparison in patients with suspected difficult airways. Minerva Anestesiol. 2013 Feb;79(2):121-9. Epub 2012 Oct 2. PMID 23032922
- [Result] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Result] Greenland KB, Edwards MJ, Hutton NJ. External auditory meatus-sternal notch relationship in adults in the sniffing position: a magnetic resonance imaging study. Br J Anaesth. 2010 Feb;104(2):268-9. doi: 10.1093/bja/aep390. No abstract available. PMID 20086071
- [Result] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Result] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Result] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341